CLINICAL TRIAL: NCT06273605
Title: Is the Use of Home-based, Dietitian-led "Egg Ladders" as a Treatment Pathway for Newly Diagnosed Infants With Immunoglobulin E (IgE) Mediated Egg Allergy Safe and Feasible? The ADAPT Program - Egg Up: A Prospective Clinical Trial
Brief Title: The Egg Up Trial - Testing a New Treatment Pathway for Infants With Newly Diagnosed Egg Allergy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 102828
Record Dates: First submitted 2024-02-01; First posted 2024-02-22 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Food Allergy; Food Allergy in Infants
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Egg Ladder (Other): An egg ladder is a form of home-based dietary advancement therapy that aims to facilitate the development of natural tolerance through the gradual introduction of egg containing foods with increasing quantity and allergenicity through different cooking processes. This intervention involves 5 steps over a 12 month period 1.baked egg, 2.well-cooked egg as an ingredient, 3. well cooked whole egg, 4. lightly cooked whole egg and 5.then raw egg.
  Interventions: Other: Egg Ladder

INTERVENTIONS:
Other: Egg Ladder — 12 month protocol of graded and gradual egg introduction

SUMMARY:
The goal of this study is to test the safety and feasibility of a change in management approach for infants with newly diagnosed egg allergy. Infants with newly diagnosed egg allergy will have egg introduced via a gradual and graded home based approach known as an "egg ladder" supervised by a dietitian. The main questions this study aims to answer are how safe and feasible are home-based dietitian-led "egg ladders" as a treatment pathway to achieve tolerance of egg for newly diagnosed infants with egg allergy.

DETAILED DESCRIPTION:
This prospective trial will evaluate the safety and feasibility of a change in practice for infants with newly diagnosed IgE-mediated egg allergy managed by the Department of Allergy and Immunology at the Royal Children's Hospital (RCH). Children <12 months of age with clinician diagnosed IgE-mediated egg allergy, who do not have a history of severe anaphylaxis to egg will be offered cautious, home-based egg introduction via a standardised 'egg ladder' protocol with dietitian support. An egg ladder is a form of dietary advancement therapy that aims to facilitate the development of natural tolerance through the gradual introduction of egg with increasing allergenicity and quantity. Although increasingly becoming widespread in clinical practice, this is yet to be evaluated in Australia via a prospective study. The HealthNuts cohort study has shown that 80% of 12-month-old infants tolerate baked egg (eg in a muffin) and 47% have naturally outgrown their egg allergy (tolerating raw egg) by 2 years of age which was 1 year from their egg allergy diagnosis.

Current practice at RCH allergy clinic for infants with egg allergy is to recommend they avoid all forms of egg until 2 years when an inpatient baked egg challenge in the form of a muffin may be offered. If passed, the children can include baked egg products at home but must avoid cooked and raw egg until a resolution challenge is offered 12 months later (cooked egg in the form of well-cooked scrambled egg). Raw egg hospital challenges are no longer offered at RCH. Review of the inpatient challenges at RCH undertaken from January - June 2023 found the median age for a baked egg challenge was 5 years and a cooked egg challenge was 4 years with a current waitlist of 1200 patients. This current model of care is prolonging the burden of food allergy management for these families for years beyond the time where resolution has likely to have occurred in the overwhelming majority. Furthermore, children are reviewed by the Allergy physician yearly if diagnosed <12 months of age and then every 2 years after that, which adds further pressure to outpatient waitlists for allergy clinics.

We will establish the safety of our 'egg ladder' protocol by collecting adverse events (AE) from baseline (egg allergy diagnosis) to final follow up (12 months after egg allergy diagnosis). The feasibility will be determined by the proportion of children who complete all stages of the egg ladder at 12 months from their diagnosis (egg allergy resolution). Barriers to completing the egg ladder protocol, parent reported quality of life and anxiety will be captured from baseline to final follow up 12 months after egg allergy diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* infants aged greater than 4 months and less than 12 months of age diagnosed by an RCH allergist with IgE- mediated egg allergy in conjunction with a positive skin prick test (SPT) or specific immunoglobulin E (sIgE) to egg white
* has a legally acceptable representative capable of understanding the informed consent document and providing consent on the participants behalf

Exclusion Criteria:

* any history of severe food induced anaphylaxis. Defined as reaction requiring 2 doses of intermuscular adrenalin
* Physician diagnosed recurrent wheeze
* Not commenced or unable to eat solid food
* prescribed beta-blocker medication

Ages: 4 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 109 (Actual)
Dates: Start 2024-04-09 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number and severity of adverse events related to baked egg ingestion (step 1) while following the home-based egg ladder protocol as collected via parent questionnaire and medical history. | 12 months
  Number, frequency and severity of adverse events as assessed by standardized predetermined criteria, related to egg ingestion (step 1 of the egg ladder - baked egg) from diagnosis until 12 months post diagnosis collected via parent questionnaire and medical history.
Number and severity of adverse events related to ingestion of well cooked egg as an ingredient (step 2) while following the home-based egg ladder protocol as collected via parent questionnaire and medical history. | 12 months
  Number, frequency and severity of adverse events as assessed by standardized predetermined criteria, related to egg ingestion (step 2 of the egg ladder - well cooked egg as an ingredient) from diagnosis until 12 months post diagnosis collected via parent questionnaire and medical history.
Number and severity of adverse events related ingestion of well cooked whole egg (step 3) while following the home-based egg ladder protocol as collected via parent questionnaire and medical history. | 12 months
  Number, frequency and severity of adverse events as assessed by standardized predetermined criteria, related to egg ingestion (step 3 of the egg ladder - well cooked whole egg) from diagnosis until 12 months post diagnosis collected via parent questionnaire and medical history.
Number and severity of adverse events related to ingestion of lightly cooked whole egg (step 4) while following the home-based egg ladder protocol as collected via parent questionnaire and medical history. | 12 months
  Number, frequency and severity of adverse events as assessed by standardized predetermined criteria, related to egg ingestion (step 4 of the egg ladder - lightly cooked whole egg) from diagnosis until 12 months post diagnosis collected via parent questionnaire and medical history.
Number and severity of adverse events related to raw egg ingestion (step 5) while following the home-based egg ladder protocol as collected via parent questionnaire and medical history. | 12 months
  Number, frequency and severity of adverse events as assessed by standardized predetermined criteria, related to egg ingestion (step 5 of the egg ladder - raw egg) from diagnosis until 12 months post diagnosis collected via parent questionnaire and medical history.
Feasibility of the home-based, egg ladder protocol to achieve egg allergy resolution 12 months from egg allergy diagnosis | 12 months
  Feasibility will be determined via clinician and parent questionnaires which will measure barriers to utilizing the egg ladder as a treatment pathway for newly diagnosed egg allergy.

SECONDARY OUTCOMES:
Change from baseline (diagnosis) in parent reported Quality of Life scores using the Food Allergy Quality of Life Questionnaire (FAQLQ-PF) to study completion (12 months from diagnosis) | Baseline, 12 months
  The Food Allergy Quality of Life Questionnaire (FAQLQ-PF) is used for assessing the Quality of Life of children with food allergies aged 0-12 years from their parents report. It gives a total mean score consisting of scores of 3 subscales: emotional impact, food anxiety, and social and dietary limitations. The FAQLQ-PF is scored using a 7-point Likert scales from 0 to 6 - a higher score indicates worse FAQL for the recall period.
Change from baseline (diagnosis) in parental anxiety scores measured using the Impairment Measure for Parental Food Allergy - Associated Anxiety and Coping Tool (IMPAACT) to study completion (12 months from diagnosis) | Baseline, 12 months
  The Impairment Measure for Parental Food Allergy-Associated Anxiety and Coping Tool (IMPAACT) is a validated 28-item self-report questionnaire for assessing food allergy-specific anxiety in the caregivers of children with food allergy. Items are completed on a 7-point Likert scale and summed to yield a total food allergy-specific anxiety score. Total IMPAACT scores range from 0 to 196 with the higher the score the greater the level of anxiety.
Heath care costs | 12 months
  Total cost of allergy related healthcare during the home-based egg ladder intervention with dietitian support from baseline (diagnosis) to study completion (12 months from diagnosis) compared to the current model of care at the Royal Children's Hospital Allergy clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Vicki McWilliam, PhD, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Murdoch Children's Research Institute (MCRI), Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set collected for this analysis of the Egg Up trial will be available six months after publication of the primary outcome. The study protocol may be obtained from the Murdoch Children's Research Institute. Prior to releasing any data the following are required: a data access agreement must be signed between relevant parties, the Egg Up trial investigators must see and approve the analysis plan describing how the data will be analyzed, there must be an agreement around appropriate acknowledgment and any additional costs involved must be covered. Should the study investigators be unavailable, this role is delegated to the Murdoch Children's Research Institute. Data will only be shared with a recognized research institute which has approved the proposed analysis plan.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication of the primary outcome
Access Criteria: Prior to releasing any data the following are required: a data access agreement must be signed between relevant parties, the Egg Up trial investigators must see and approve the analysis plan describing how the data will be analyzed, there must be an agreement around appropriate acknowledgment and any additional costs involved must be covered.

REFERENCES:
- [Background] McAdams SA, Cordeiro ML. Simple selected ion monitoring capillary gas chromatographic-mass spectrometric method for the determination of cotinine in serum, urine and oral samples. J Chromatogr. 1993 May 19;615(1):148-53. doi: 10.1016/0378-4347(93)80301-j. PMID 8340453
- [Background] Bettocchi S, Di Vagno G, Cormio G, Selvaggi L. Intra-abdominal spread of malignant cells following hysteroscopy. Gynecol Oncol. 1997 Jul;66(1):165-6. doi: 10.1006/gyno.1997.4654. No abstract available. PMID 9234941
- [Background] Koplin JJ, Wake M, Dharmage SC, Matheson M, Tang ML, Gurrin LC, Dwyer T, Peters RL, Prescott S, Ponsonby AL, Lowe AJ, Allen KJ; HealthNuts study group. Cohort Profile: The HealthNuts Study: Population prevalence and environmental/genetic predictors of food allergy. Int J Epidemiol. 2015 Aug;44(4):1161-71. doi: 10.1093/ije/dyu261. Epub 2015 Jan 21. PMID 25613427
- [Background] Leech SC, Ewan PW, Skypala IJ, Brathwaite N, Erlewyn-Lajeunesse M, Heath S, Ball H, James P, Murphy K, Clark AT. BSACI 2021 guideline for the management of egg allergy. Clin Exp Allergy. 2021 Oct;51(10):1262-1278. doi: 10.1111/cea.14009. PMID 34586690